CLINICAL TRIAL: NCT01207817
Title: Effect of Ambient Light on the Parameters of the Pupillary Light Reflex
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Lawrence Chin, MD, UMDNJ
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0120090181
Record Dates: First submitted 2010-01-25; First posted 2010-09-23 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Volunteers
Keywords: a light flash in each eye for a total of 48 measurements

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no condition: no condition - healthy volunteers
  Interventions: Other: Pupillometry

INTERVENTIONS:
Other: Pupillometry — Pupillometry readings will be taken at low, intermediate and high ambient light

SUMMARY:
The purpose of this study is to determine the effects of varying luminescent levels on the pupillary response.

DETAILED DESCRIPTION:
Evaluation of the pupillary response is an underemphasized aspect of the assessment of visual function. The pupillary light reflex is one of the few objective indicators of afferent input from the retina and optic nerve. Since the pupillary light reflex is processed through the retina, it may be used to assess visual integrity (1). Pupillometry is a reliable technology capable of providing repetitive data on quantitative pupillary function in states of health and disease (2). Amplitude, latency, maximum constriction velocity, mean constriction velocity, and dilation velocity are measured using the Neuroleptics pupillometer. The effects of varying levels of ambient light on these parameters of the pupillary response have not been extensively studied. The purpose of this investigation is to determine the effects of varying luminescent levels on the pupillary response.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* recent bout of conjunctivitis or infection in the eye recent eye surgery seizure disorder unable to lie flat for 30 minutes known history of eye disease which cannot be corrected with lenses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volinteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
pupillary light reflex: amplitude, latency, maximum constriction velocity, mean constriction velocity and dilation velocity during different levels of ambient light | Pupillometry readings will be taken at 3 potential light readings low light, intermediate light and high ambient light. A total of 48 readings will be done. All parameters will be done at one sitting and will take approximately 45 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence W Chinn, MD, Principal Investigator — UMDNJ-NJMS
Locations (1):
- UMDNJ-University Hospital, Newark, New Jersey, United States